CLINICAL TRIAL: NCT01048112
Title: Campylobacter Jejuni Challenge Model Development: Assessment of Homologous Protection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: United States Army Medical Materiel Development Activity (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Beth Kirkpatrick, MD, University of Vermont
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRMS 10-086; NMRC 2009.0017 (Other: NMRC IRB)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Campylobacter Infections
Keywords: campylobacter; gastroenteritis; challenge models
MeSH Terms: conditions — Campylobacter Infections; Gastroenteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repeated dose group (Experimental): Will receive one dose of Campylobacter jejuni strain CG8421 at day 0 and a second dose at approximately day 98.
  Interventions: Biological: Campylobacter jejuni strain CG8421
- Single dose group (Active Comparator): Will receive one dose of Campylobacter jejuni strain CG8421
  Interventions: Biological: Campylobacter jejuni strain CG8421

INTERVENTIONS:
Biological: Campylobacter jejuni strain CG8421 — Single oral dose of Campylobacter jejuni strain CG8421 in sodium bicarbonate buffer

SUMMARY:
The goal of this research is to continue to develop a model of infection with Campylobacter jejuni, a bacterium that causes food and water-borne disease (mainly diarrhea). The objectives are to 1) determine if healthy subjects develop short-term (<6 month) protection to reinfection with C. jejuni; and 2) characterize the immune responses to C. jejuni infection. Information obtained will be used in development of a vaccine against Campylobacter infections.

Volunteers will be screened for eligibility within 60 days prior to enrollment. Screening will include obtaining informed consent prior to any study procedure. This will be followed by medical history, physical examination, review of current medications, blood samples for safety labs (WBC, Hct, Hgb, platelet count; chemistry panel; screening for HIV, HLA-B27, HBV, and HCV); urine pregnancy testing for females. Stool will be tested for infection.

Eligible volunteers will be enrolled in the study and admitted to the GCRC on Day -1. They will drink a measured dose of C. jejuni on Day 0, and followed for approximately 9 inpatient days, during which time the investigators expect at least 75% to develop a diarrheal illness, which will be promptly treated with replacement fluids (oral or IV, as indicated) and antibiotics. During the inpatient period, subjects will be assessed for any adverse events, and blood and stool specimens will be analyzed for markers of infection and markers of immune response. Subjects must have resolved or resolving symptoms and two negative stool cultures ≥12 hours apart to be eligible for discharge, and will be seen in outpatient follow-up at 21, 28, 35, 60, and 90 days for additional AE assessments and blood and stool analysis.

Eight subjects will return for redosing approximately 98 days after the initial dose, with the same inpatient and outpatient follow-up as above. Few or none should develop a diarrheal illness. Four naïve (previously unexposed) subjects will also receive the dose on Day 98 to confirm a 75% illness rate with this dose. They will be followed as the initial group was. All participants will be assessed by phone 6 months after the final dose they received.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age, inclusive.
* General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by principal investigator or principal investigator in consultation with the medical monitor and sponsor.
* Demonstrate comprehension of the protocol procedures and knowledge of Campylobacter illness by passing a written examination (pass grade ≥ 70%)
* Willing to participate after informed consent obtained.
* Available for all planned follow-up visits, and remain available for medical interview/physical exam and monitoring for 90 days post-challenge (last challenge received), and a final telephone interview 180 days post-challenge.
* Negative urine pregnancy test at screening and a negative urine pregnancy test on the day of admittance to the inpatient phase for all female subjects. In addition, female subjects will be advised of the need for an effective means of birth control during the entire study period.

Exclusion Criteria:

* Presence of a significant medical condition (e.g., psychiatric conditions; gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis, inflammatory bowel disease, irritable bowel syndrome; alcohol or illicit drug abuse/dependency), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
* Immunosuppressive illness, IgA deficiency (below the normal limits), or H2 antihistamine use within 48 h of admission or during inpatient period.
* Positive serology results for HIV, HBsAg, or HCV antibodies.
* Significant abnormalities in screening lab hematology, serum chemistry, as determined by PI or PI in consultation with the medical monitor and sponsor.
* Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding receipt of the challenge inoculum or planned use during the active study period.
* Nursing mother on the day of admittance to the inpatient phase for all female subjects.
* Are not capable of fully informed consent (e.g., cannot read or write English)
* Personal or documented family history of an inflammatory arthritis such as reactive arthritis, Reiter's syndrome, ankylosing spondylitis, rheumatoid arthritis, or Guillain-Barré syndrome (would not include osteoarthritis or vague history of arthritis in a relative late in adulthood).
* Evidence of neurologic abnormalities (specifically extremity weakness, abnormal deep tendon reflexes, symmetric sensory abnormalities - vibratory, light touch, and proprioception).
* Evidence of inflammatory arthritis on exam and/or HLA-B27 positive (flow cytometry).
* Allergy or prior intolerance to any of the following antibiotics: azithromycin, fluoroquinolones, or penicillin.
* Fewer than 3 stools per week or more than 3 stools per day as the usual frequency, loose or liquid stools other than on an occasional basis.
* Regular use of laxatives or any agent that increases gastric pH (regular defined as at least weekly).
* Have household contacts who are <2 years old or >80 years old or infirmed or immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease).
* Employment as either a health care worker with direct patient care, in a daycare center (for children or the elderly), or working directly with food.
* History of microbiologically confirmed Campylobacter infection
* Immunologic evidence of Campylobacter exposure
* Individuals who have traveled to countries with high Campylobacter rates within the past two years and who experienced an episode of diarrhea during or within 1 week of returning from their trip.
* And others

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Development of campylobacteriosis in response to a dose of Campylobacter jejuni strain CG8421 | 10 days
Immunologic responses to dosing with Campylobacter jejuni strain CG8421 | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth Kirkpatrick, MD, Principal Investigator — University of Vermont; David Tribble, MD, Principal Investigator — Navy Medical Research Center
Locations (2):
- United States (2):
  - Navy Medical Research Center, Silver Spring, Maryland
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Kirkpatrick BD, Lyon CE, Porter CK, Maue AC, Guerry P, Pierce KK, Carmolli MP, Riddle MS, Larsson CJ, Hawk D, Dill EA, Fingar A, Poly F, Fimlaid KA, Hoq F, Tribble DR. Lack of homologous protection against Campylobacter jejuni CG8421 in a human challenge model. Clin Infect Dis. 2013 Oct;57(8):1106-13. doi: 10.1093/cid/cit454. Epub 2013 Jul 9. PMID 23840001
- See also: UVM Vaccine Testing Center — http://www.med.uvm.edu/Medicine/ID/TB3+CL+BL+3I.asp?SiteAreaID=616